CLINICAL TRIAL: NCT02627430
Title: A Phase 1 Study of PARP Inhibitor BMN 673 and HSP90 Inhibitor AT13387 for Treatment of Advanced Solid Tumors With Expansion in Patients With Recurrent Epithelial Ovarian, Fallopian Tube, Peritoneal Cancer or Recurrent Triple-Negative Breast Cancer
Brief Title: Talazoparib and HSP90 Inhibitor AT13387 in Treating Patients With Metastatic Advanced Solid Tumor or Recurrent Ovarian, Fallopian Tube, Primary Peritoneal, or Triple Negative Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Other - Protocol moved to Withdrawn
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-02063; NCI-2015-02063 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9896 (Other: Dana-Farber - Harvard Cancer Center LAO); 9896 (Other: CTEP); P30CA006516 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2015-12-09; First posted 2015-12-11 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Adult Solid Neoplasm; Estrogen Receptor Negative; Fallopian Tube Serous Neoplasm; HER2/Neu Negative; Ovarian Serous Adenocarcinoma; Ovarian Serous Tumor; Primary Peritoneal Serous Adenocarcinoma; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Triple Negative Breast Neoplasms | interventions — (2,4-dihydroxy-5-isopropylphenyl)-(5-(4-methylpiperazin-1-ylmethyl)-1,3-dihydroisoindol-2-yl)methanone; talazoparib

ARMS (1):
- Treatment (talazoparib and Hsp90 inhibitor AT13387) (Experimental): Patients receive talazoparib PO QD on days 1-7 (course 0). Beginning in course 1, patients receive talazoparib PO QD on days 1-28 and HSP90 inhibitor AT13387 IV over 1 hour on days 1, 2, 8, 9, 15, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Hsp90 Inhibitor AT13387; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Talazoparib

INTERVENTIONS:
Drug: Hsp90 Inhibitor AT13387 — Given IV
  Other Names: AT13387
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Talazoparib — Given PO
  Other Names: BMN 673; BMN-673

SUMMARY:
This phase I trial studies the side effects and best dose of talazoparib and heat shock protein (HSP)90 inhibitor AT13387 when given together in treating patients with solid tumors that have spread to other places in the body (metastatic) or ovarian, fallopian tube, primary peritoneal, or hormone negative breast cancer that have come back after a period of improvement (recurrent). Talazoparib and HSp90 inhibitor AT13387 may stop the growth of tumor cells by blocking some enzymes that are need for cell growth. HSp90 inhibitor AT1338 may also help talazoparib work better by making tumor cells more sensitive to the drug.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTDs) of BMN673 (talazoparib) and AT13387 (HSP90 Inhibitor AT13387) administered in combination in patients with advanced solid tumors.

SECONDARY OBJECTIVES:

I. To identify the dose-limiting toxicity (DLT) and other toxicities associated with BMN673 and AT13387 administered in combination as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v) 4.0.

II. To determine the recommended phase 2 doses (RP2D) of the combination of BMN673 and AT13387.

III. To determine the plasma pharmacokinetics of BMN673 and AT13387. IV. To document anti-tumor activity of the combination of BMN673 and AT13387 as assessed by (Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and progression free survival (PFS).

OUTLINE: This is a dose-escalation study.

Patients receive talazoparib orally (PO) once daily (QD) on days 1-7 (course 0). Beginning in course 1, patients receive talazoparib PO QD on days 1-28 and HSP90 inhibitor AT13387 intravenously (IV) over 1 hour on days 1, 2, 8, 9, 15, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* For the dose escalation cohort, patients must have histologically or cytologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* For the dose expansion cohort, participants must have histologically or cytologically confirmed diagnosis of either: i) ovarian, fallopian tube, or primary peritoneal cancer of high grade serous histology which has recurred despite standard therapy or ii) triple-negative breast cancer which has recurred despite standard therapy
* There is no line limit for the dose escalation cohort and the dose expansion cohort
* For the dose expansion cohort, patients with ovarian, fallopian tube or primary peritoneal cancer must have platinum resistant disease defined as progression within 6 months after last platinum regimen; platinum refractory disease is allowed
* For the dose expansion cohort, patients with triple-negative breast cancer may not be breast cancer 1/2 (BRCA1/2) germline mutation carriers
* There must be availability of a formalin-fixed, paraffin-embedded tumor specimen with adequate viable tumor tissue
* Eastern Cooperative Oncology Group (ECOG) performance status < 2 (Karnofsky > 60)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) = < 2.5 × institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Left ventricular ejection fraction > 50% on echocardiography or multigated acquisition (ECHO/MUGA) scan
* Corrected QT (QTc) =< 450 ms
* Any clinically significant electrolyte imbalance, particularly hypokalemia and hypomagnesemia, should be corrected before treatment
* Have undergone clearance after baseline ophthalmologic exam (at least fundoscopic exam, visual acuity, intraocular pressure, assessment of visual fields and measurement of color vision)
* For the expansion cohort only: measurable disease by RECIST v1.1 with at least one measurable target lesion
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of BMN 673 and/or AT13387 administration
* Patients must be able to swallow pills and have no significant impairment in gastrointestinal absorption
* Three biopsies, one pretreatment, one after BMN673 alone and one after one of the combinations of BMN673/AT13387 will be voluntary in the expansion and dose escalation cohorts; however, biopsies will be required in at least 8 patients of the 20 patients to be enrolled in the expansion cohort
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* All acute, clinically significant treatment-related toxicity from prior therapy, except for alopecia, must have resolved to grade =< 1
* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BMN 673 and AT13387 used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with BMN 673 or AT13387
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Known history of QT/QTc prolongation or torsades de pointes (TdP); patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing torsades de pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
MTD based on the dose-limiting toxicity based on the National Cancer Institute (NCI) CTCAE v. 4.0 | 35 days
  DLT defined as non-hematologic and hematologic toxicities experienced during course 0 and the first course (i.e. first 4 weeks) of treatment.

SECONDARY OUTCOMES:
Incidence of adverse events as assessed by NCI CTCAE v. 4.0 | 30 days post-treatment
Pharmacokinetic (PK) parameters of talazoparib and HSP90 inhibitor AT13387 | Baseline, at 1, 2, 4 and 8 hours of day 1 (course 0), baseline of days 1, 8, and 15 of course 1, and at 1, 2, 4, and 8 hours post-dosing on day 8 and 15 of course 1
  Pearson correlation coefficients, presented with 95% confidence intervals, will be used to investigate the association of the percent change heat shock protein 90 and poly(adenosine diphosphate-ribose) polymerase 1 activities with PK parameters, including maximum concentration observed and area under the curve.

OTHER OUTCOMES:
Change in BRCA1 foci expression in tumor tissue via IHC | Baseline to day 15 of course 1
  Paired t-tests will be used to compare BRCA1 foci formation following BMN673/AT13387.
Change in BRCA1 foci expression in tumor tissue via immunohistochmestry (IHC) | Baseline to day 7 of course 0
  Paired t-tests will be used to compare BRCA1 foci formation following BMN673.
Change in heat shock protein 70 (HSPT70) expression | Day 7 (course 0) to day 15 (course 1)
  Changes in parameters of HSP70 activities that occur post-treatment will be summarized using descriptive statistics.
Change in RAD51 foci expression in tumor tissue via IHC | Baseline to day 15 of course 1
  Paired t-tests will be used to compare RAD51 foci formation following BMN673/AT13387.
Change in RAD51 recombinase (RAD51) foci expression in tumor tissue via IHC | Baseline to day 7 of course 0
  Paired t-tests will be used to compare RAD51 foci formation following BMN673.

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Konstantinopoulos, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO